CLINICAL TRIAL: NCT05590585
Title: An Open-Label Single-Arm Study of Dupilumab in Adolescent and Adult Skin of Color Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Dupilumab in Adolescent and Adult Skin of Color Participants: Open-label Moderate-to-severe Eczema Trial
Acronym: DISCOVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-2217
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Moderate-to-Severe Atopic Dermatitis; Atopic Eczema
Keywords: Eczematous Lesions; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — dupilumab; Emollients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dupilumab (Experimental): Adolescents and adults will receive 1 of 2 dose regimens based on age and body weight
  Interventions: Drug: dupilumab; Other: Topical emollient (moisturizer)

INTERVENTIONS:
Drug: dupilumab — Administered by subcutaneous (SC) injection once every 2 weeks (Q2W) following a loading dose
  Other Names: Dupixent®; R668; SAR231893
Other: Topical emollient (moisturizer) — Moisturizer should be applied twice daily, as per physician's recommendation, as defined in protocol.

SUMMARY:
The study is focused on skin of color participants who have moderate-to-severe atopic dermatitis. Atopic dermatitis, also referred to as eczema, is a condition that causes the skin to become itchy, dry, and cracked.

From the previous studies on the study drug, it is seen that the study drug has an acceptable safety and effectiveness in participants with atopic dermatitis.

The aim of this study is to get additional information on the safety and effectiveness of the study drug, particularly the information on aspects of atopic dermatitis in skin of color participants.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in your blood at different times
* How much the study drug improves quality of life and mental health

ELIGIBILITY:
Key Inclusion Criteria:

1. Skin of color, defined as Fitzpatrick skin type ≥4 at screening visit
2. Diagnosis of moderate-to-severe atopic dermatitis (AD) that cannot be adequately controlled with topical AD medications, as defined in protocol
3. Has applied a stable dose of topical emollient (moisturizer) twice daily as per physician recommendation starting at screening visit

Key Exclusion Criteria:

1. Self-reported Caucasian or White race
2. Adolescent body weight less than 30 kg at screening
3. Prior use of dupilumab within 6 months of screening
4. Concomitant skin diseases or other pigmentary disorder that could confound AD assessments
5. Current or prior use, within 12 weeks before the screening visit, of phototherapy or tanning beds
6. Active helminthic infections; suspected or high risk of helminthic infection, unless clinical and (if necessary) laboratory assessments have ruled out active infection before baseline
7. Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 7 days prior to baseline
8. Planned or anticipated use of any prohibited medications and procedures, as defined in protocol
9. Has received a COVID-19 vaccination within 1 week of planned start of study medication or for which the planned COVID-19 vaccinations would not be completed 1 week prior to start of study drug

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (30):
- United States (30):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - The University Of Alabama At Birmingham, Birmingham, Alabama
  - C2 Research Center, LLC, Montgomery, Alabama
  - Center for Dermatology Clinical Research, inc., Fremont, California
  - UCSD/ Rady Children's Hospital, San Diego, California
  - UCSF, San Francisco, California
  - SF Research Institute, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Skin and Cancer Associates, LLP, Miami, Florida
  - Century Research LLC, Miami, Florida
  - Advanced Medical Research PC, Atlanta, Georgia
  - Atlanta Biomedical Clinical Research LLC, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Callender Dermatology and Cosmetic Center, Glenn Dale, Maryland
  - Dermatology and Skin Cancer Specialists, LLC dba US Dermatology Partners, Rockville, Maryland
  - Wayne State University Physician Group Dermatology, Dearborn, Michigan
  - Revival Research Institute , LLC, Troy, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Rao Dermatology, Atlantic Highlands, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - NYC Health + Hospital , Elmhurst Hospital Center, Elmhurst, New York
  - Markowitz Medical, New York, New York
  - Philip Fried, MD PLLC, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - National Allergy and Asthma Research, LLC., North Charleston, South Carolina
  - Center for Clinical Studies, LTD.LLP, Houston, Texas
  - Heights Dermatology & Aesthetic Center - Heights Location, Houston, Texas
  - RFSA Dermatology, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at a total of 30 sites located in the United States. A total of 166 participants were screened for the study, of which 124 were enrolled and were treated with dupilumab.
Groups:
- Dupilumab: Participants received dupilumab by subcutaneous (SC) injection once every 2 weeks (Q2W) for 24 weeks following a loading dose based on age and body weight.
Period: Overall Study
Arm/Group | Dupilumab
Started | 124
Received at Least 1 Dose of Dupilumab | 124
Completed | 120
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who were enrolled in the study and had at least 1 post-baseline efficacy assessment.
Groups:
- Dupilumab: Participants received dupilumab by SC injection Q2W for 24 weeks following a loading dose based on age and body weight.
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3
  Race: Black or African American | 98
  Race: Asian | 13
  Race: American Indian or Alaska Native | 3
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Other | 3

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Score 0 to 1
Description: IGA is an assessment scale used to determine severity of atopic dermatitis (AD) and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). Percentage of participants with IGA "0" or "1" are reported at each visit.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 0.9
  Week 4: number analyzed (Participants) | 117
  Week 4 | 6.8
  Week 8: number analyzed (Participants) | 113
  Week 8 | 15.9
  Week 12: number analyzed (Participants) | 108
  Week 12 | 25.9
  Week 16: number analyzed (Participants) | 108
  Week 16 | 35.2
  Week 20: number analyzed (Participants) | 97
  Week 20 | 45.4
  Week 24: number analyzed (Participants) | 100
  Week 24 | 44.0

2. Secondary Outcome: Percent Change From Baseline in EASI Score
Description: The Eczema Area and Severity Index (EASI) score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percent change
  Week 2: number analyzed (Participants) | 116
  Week 2 | -25.929 (29.782)
  Week 4: number analyzed (Participants) | 117
  Week 4 | -46.092 (30.000)
  Week 8: number analyzed (Participants) | 113
  Week 8 | -67.270 (25.689)
  Week 12: number analyzed (Participants) | 108
  Week 12 | -70.999 (25.798)
  Week 16: number analyzed (Participants) | 108
  Week 16 | -73.276 (32.975)
  Week 20: number analyzed (Participants) | 97
  Week 20 | -79.185 (23.612)
  Week 24: number analyzed (Participants) | 100
  Week 24 | -79.941 (25.634)

3. Secondary Outcome: Change From Baseline in EASI Score
Description: as for outcome 2
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
score on scale
  Week 2: number analyzed (Participants) | 116
  Week 2 | -7.105 (7.504)
  Week 4: number analyzed (Participants) | 117
  Week 4 | -12.097 (9.338)
  Week 8: number analyzed (Participants) | 113
  Week 8 | -17.779 (10.178)
  Week 12: number analyzed (Participants) | 108
  Week 12 | -18.475 (9.768)
  Week 16: number analyzed (Participants) | 108
  Week 16 | -19.460 (11.663)
  Week 20: number analyzed (Participants) | 97
  Week 20 | -20.985 (11.249)
  Week 24: number analyzed (Participants) | 100
  Week 24 | -20.980 (11.071)

4. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in EASI Score (EASI-50)
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50 responders were the participants who achieved ≥50% overall improvement in EASI score from baseline to the given time point.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 17.2
  Week 4: number analyzed (Participants) | 117
  Week 4 | 47.9
  Week 8: number analyzed (Participants) | 113
  Week 8 | 77.9
  Week 12: number analyzed (Participants) | 108
  Week 12 | 84.3
  Week 16: number analyzed (Participants) | 108
  Week 16 | 84.3
  Week 20: number analyzed (Participants) | 97
  Week 20 | 89.7
  Week 24: number analyzed (Participants) | 100
  Week 24 | 89.0

5. Secondary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in EASI Score (EASI-75)
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to the given time point.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 3.4
  Week 4: number analyzed (Participants) | 117
  Week 4 | 23.1
  Week 8: number analyzed (Participants) | 113
  Week 8 | 50.4
  Week 12: number analyzed (Participants) | 108
  Week 12 | 56.5
  Week 16: number analyzed (Participants) | 108
  Week 16 | 63.9
  Week 20: number analyzed (Participants) | 97
  Week 20 | 74.2
  Week 24: number analyzed (Participants) | 100
  Week 24 | 76.0

6. Secondary Outcome: Percentage of Participants With ≥90% Reduction From Baseline in EASI Score (EASI-90)
Description: The EASI score was used to measure the severity and extent of AD and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-90 responders were the participants who achieved ≥90% overall improvement in EASI score from baseline to the given time point.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 116
  Week 2 | 0.9
  Week 4: number analyzed (Participants) | 117
  Week 4 | 5.1
  Week 8: number analyzed (Participants) | 113
  Week 8 | 15.0
  Week 12: number analyzed (Participants) | 108
  Week 12 | 27.8
  Week 16: number analyzed (Participants) | 108
  Week 16 | 38.9
  Week 20: number analyzed (Participants) | 97
  Week 20 | 41.2
  Week 24: number analyzed (Participants) | 100
  Week 24 | 42.0

7. Secondary Outcome: Percent Change From Baseline in Total Scoring Atopic Dermatitis (SCORAD) Score
Description: The SCORAD index is a clinical tool for assessing the severity of atopic dermatitis. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percent change
  Week 2: number analyzed (Participants) | 110
  Week 2 | -18.5 (17.8)
  Week 4: number analyzed (Participants) | 111
  Week 4 | -30.2 (22.6)
  Week 8: number analyzed (Participants) | 107
  Week 8 | -44.4 (22.8)
  Week 12: number analyzed (Participants) | 102
  Week 12 | -50.5 (23.0)
  Week 16: number analyzed (Participants) | 102
  Week 16 | -53.2 (26.0)
  Week 20: number analyzed (Participants) | 91
  Week 20 | -55.6 (24.3)
  Week 24: number analyzed (Participants) | 94
  Week 24 | -59.3 (26.0)

8. Secondary Outcome: Percentage of Participants With ≥50% Reduction From Baseline in SCORAD Score (SCORAD-50)
Description: SCORAD index is a clinical tool for assessing the severity of atopic dermatitis. Extent and intensity of eczema as well as subjective signs insomnia, etc.) were assessed and scored. Total score ranged from 0 (absent disease) to 103 (severe disease). A decrease in score indicated improvement.
  SCORAD-50 was defined as ≥50% reduction from baseline in SCORAD score.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 110
  Week 2 | 9.1
  Week 4: number analyzed (Participants) | 111
  Week 4 | 16.2
  Week 8: number analyzed (Participants) | 107
  Week 8 | 39.3
  Week 12: number analyzed (Participants) | 102
  Week 12 | 52.9
  Week 16: number analyzed (Participants) | 102
  Week 16 | 59.8
  Week 20: number analyzed (Participants) | 91
  Week 20 | 68.1
  Week 24: number analyzed (Participants) | 94
  Week 24 | 70.2

9. Secondary Outcome: Percentage of Participants With Improvement (Reduction) From Baseline of Weekly Average of Daily Peak Pruritus (PP) Numerical Rating Scale (NRS) Score ≥3
Description: Peak Pruritus NRS is an assessment tool used by participants to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" For post-baseline NRS, the mean weekly NRS was calculated as the prorated average of the reported daily NRS within the week. A decrease in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 119
  Week 2 | 14.3
  Week 4: number analyzed (Participants) | 117
  Week 4 | 31.6
  Week 8: number analyzed (Participants) | 114
  Week 8 | 48.2
  Week 12: number analyzed (Participants) | 108
  Week 12 | 54.6
  Week 16: number analyzed (Participants) | 108
  Week 16 | 64.8
  Week 20: number analyzed (Participants) | 103
  Week 20 | 68.0
  Week 24: number analyzed (Participants) | 93
  Week 24 | 65.6

10. Secondary Outcome: Percentage of Participants With Improvement (Reduction) From Baseline of Weekly Average of Daily PP NRS Score ≥4
Description: as for outcome 9
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
percentage of participants
  Week 2: number analyzed (Participants) | 119
  Week 2 | 8.4
  Week 4: number analyzed (Participants) | 117
  Week 4 | 19.7
  Week 8: number analyzed (Participants) | 114
  Week 8 | 32.5
  Week 12: number analyzed (Participants) | 108
  Week 12 | 38.9
  Week 16: number analyzed (Participants) | 108
  Week 16 | 44.4
  Week 20: number analyzed (Participants) | 103
  Week 20 | 47.6
  Week 24: number analyzed (Participants) | 93
  Week 24 | 52.7

11. Secondary Outcome: Percent Change From Baseline in Weekly Average of Daily PP NRS Score
Description: as for outcome 9
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Dupilumab
Number analyzed (Participants) | 119
Percentage of change
  Week 2 | -16.253 (25.364)
  Week 4: number analyzed (Participants) | 117
  Week 4 | -28.672 (28.427)
  Week 8: number analyzed (Participants) | 114
  Week 8 | -41.010 (33.346)
  Week 12: number analyzed (Participants) | 108
  Week 12 | -45.944 (31.358)
  Week 16: number analyzed (Participants) | 108
  Week 16 | -52.706 (30.812)
  Week 20: number analyzed (Participants) | 103
  Week 20 | -54.138 (28.698)
  Week 24: number analyzed (Participants) | 93
  Week 24 | -56.337 (31.036)

12. Secondary Outcome: Change From Baseline in Weekly Average of Daily PP NRS Score
Description: Peak Pruritus NRS is an assessment tool used by subjects to report intensity of pruritus (itch) during a 24-hour recall period. Participants were asked the following question: For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable,' how would you rate your itch at the worst moment during the previous 24 hours?" For post-baseline NRS, the mean weekly NRS was calculated as the prorated average of the reported daily NRS within the week. A decrease in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 119
score on a scale
  Week 2 | -1.234 (1.663)
  Week 4: number analyzed (Participants) | 117
  Week 4 | -2.058 (2.021)
  Week 8: number analyzed (Participants) | 114
  Week 8 | -2.939 (2.379)
  Week 12: number analyzed (Participants) | 108
  Week 12 | -3.237 (2.266)
  Week 16: number analyzed (Participants) | 108
  Week 16 | -3.741 (2.369)
  Week 20: number analyzed (Participants) | 103
  Week 20 | -3.823 (2.184)
  Week 24: number analyzed (Participants) | 93
  Week 24 | -3.981 (2.326)

13. Secondary Outcome: Percent Change From Baseline in Percent Body Surface Area (BSA)
Description: BSA affected by AD was assessed for each section of the body using the rule of nines (the possible highest score for each region was: head and neck [9%], interior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). BSA was reported as a percentage of all major body sections combined.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Dupilumab
Number analyzed (Participants) | 120
Percentage of change
  Week 2: number analyzed (Participants) | 116
  Week 2 | -17.91 (24.92)
  Week 4: number analyzed (Participants) | 117
  Week 4 | -31.07 (31.06)
  Week 8: number analyzed (Participants) | 113
  Week 8 | -53.09 (30.67)
  Week 12: number analyzed (Participants) | 108
  Week 12 | -60.04 (31.45)
  Week 16: number analyzed (Participants) | 108
  Week 16 | -64.65 (32.79)
  Week 20: number analyzed (Participants) | 97
  Week 20 | -71.03 (28.50)
  Week 24: number analyzed (Participants) | 100
  Week 24 | -73.69 (28.31)

14. Secondary Outcome: Change From Baseline in Health-related Quality of Life (QOL) as Measured by Dermatology Life Quality Index (DLQI; Age ≥16) Score
Description: DLQI is a 10-item, validated questionnaire to assess the impact of AD disease symptoms and treatment on QOL; over the past week, with an overall scoring of 0 (no effect on QoL) to 30 (extremely large effect on QoL). A decrease in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 94
score on a scale
  Week 2: number analyzed (Participants) | 91
  Week 2 | -4.5 (5.4)
  Week 4: number analyzed (Participants) | 91
  Week 4 | -5.6 (7.1)
  Week 8: number analyzed (Participants) | 88
  Week 8 | -6.7 (6.5)
  Week 12: number analyzed (Participants) | 81
  Week 12 | -7.6 (5.7)
  Week 16: number analyzed (Participants) | 84
  Week 16 | -7.6 (6.7)
  Week 20: number analyzed (Participants) | 77
  Week 20 | -8.5 (6.5)
  Week 24: number analyzed (Participants) | 71
  Week 24 | -8.3 (7.1)

15. Secondary Outcome: Change From Baseline in Health-related QOL as Measured by Children's Dermatology Life Quality Index (CDLQI; Age <16) Score
Description: CDLQI is a 10-item, validated questionnaire to assess the impact of AD disease symptoms and treatment on quality of life (QOL); over the past week, with an overall scoring of 0 (no effect on QoL) to 30 (extremely large effect on QoL) in children. A decrease in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 10
score on a scale
  Week 2 | -4.2 (5.4)
  Week 4: number analyzed (Participants) | 9
  Week 4 | -5.0 (5.2)
  Week 8: number analyzed (Participants) | 8
  Week 8 | -5.1 (4.2)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -6.3 (7.0)
  Week 16: number analyzed (Participants) | 8
  Week 16 | -8.5 (5.6)
  Week 20: number analyzed (Participants) | 7
  Week 20 | -8.6 (5.4)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -7.8 (5.5)

16. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Total Score
Description: POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (Higher score indicative of more severe symptoms). Total score was an average of the disease symptoms assessed. A decrease in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 104
score on a scale
  Week 2: number analyzed (Participants) | 101
  Week 2 | -5.6 (6.0)
  Week 4: number analyzed (Participants) | 100
  Week 4 | -8.3 (6.6)
  Week 8: number analyzed (Participants) | 96
  Week 8 | -10.3 (6.5)
  Week 12: number analyzed (Participants) | 90
  Week 12 | -11.0 (6.3)
  Week 16: number analyzed (Participants) | 92
  Week 16 | -11.2 (7.0)
  Week 20: number analyzed (Participants) | 84
  Week 20 | -11.3 (7.0)
  Week 24: number analyzed (Participants) | 80
  Week 24 | -11.5 (7.0)

17. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Total Score
Description: The Hospital Anxiety and Depression Scale (HADS) is a screening tool designed to assess anxiety and depression. The scale consists of 14 items, divided into two subscales: Anxiety (HADS-A): 7 items; Depression (HADS-D): 7 items. The range of the total score is 0-42 (sum of HADS-A and HADS-D), with higher score indicating more severe overall psychological distress. The two subscales can be reported separately, each with a score range of 0-21, with higher score indicating more severe symptoms of anxiety or depression. A decrease in either the total score or a subscale score indicates improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 104
score on a scale
  Week 2: number analyzed (Participants) | 101
  Week 2 | -1.8 (5.0)
  Week 4: number analyzed (Participants) | 100
  Week 4 | -2.3 (5.5)
  Week 8: number analyzed (Participants) | 96
  Week 8 | -2.8 (5.6)
  Week 12: number analyzed (Participants) | 89
  Week 12 | -3.7 (5.5)
  Week 16: number analyzed (Participants) | 92
  Week 16 | -3.4 (5.8)
  Week 20: number analyzed (Participants) | 84
  Week 20 | -3.4 (6.1)
  Week 24: number analyzed (Participants) | 80
  Week 24 | -3.2 (6.3)

18. Secondary Outcome: Change From Baseline in Skin Pain NRS (SP NRS) Score
Description: SP NRS Scale is an assessment tool used to report the intensity of a participant's pain. Participants selected the number between 0 and 10 that fit best to their worst pain intensity over the past 24 hours (0 = no pain and 10 = the worst pain imaginable). A decrease in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 104
score on a scale
  Week 2: number analyzed (Participants) | 101
  Week 2 | -2.3 (3.6)
  Week 4: number analyzed (Participants) | 100
  Week 4 | -2.6 (4.0)
  Week 8: number analyzed (Participants) | 96
  Week 8 | -3.2 (3.5)
  Week 12: number analyzed (Participants) | 90
  Week 12 | -3.3 (3.5)
  Week 16: number analyzed (Participants) | 92
  Week 16 | -3.0 (3.4)
  Week 20: number analyzed (Participants) | 84
  Week 20 | -3.0 (3.2)
  Week 24: number analyzed (Participants) | 80
  Week 24 | -2.9 (3.5)

19. Secondary Outcome: Change From Baseline in Weekly Average Sleep Quality NRS Score
Description: Sleep Quality NRS is an 11-point scale (0 to 10) in which 0 indicated worst possible sleep while 10 indicated best possible sleep. An increase in score indicated improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dupilumab
Number analyzed (Participants) | 119
score on a scale
  Week 2: number analyzed (Participants) | 80
  Week 2 | 0.473 (1.565)
  Week 4: number analyzed (Participants) | 84
  Week 4 | 0.910 (1.937)
  Week 8: number analyzed (Participants) | 84
  Week 8 | 1.204 (2.459)
  Week 12: number analyzed (Participants) | 72
  Week 12 | 1.281 (2.173)
  Week 16: number analyzed (Participants) | 72
  Week 16 | 1.239 (2.097)
  Week 20: number analyzed (Participants) | 67
  Week 20 | 1.045 (2.631)
  Week 24: number analyzed (Participants) | 58
  Week 24 | 1.210 (2.696)

20. Secondary Outcome: Percentage of Participants With Patient Global Impression of Disease (PGID) Response as No Symptoms
Description: PGID is a single 1-item questionnaire designed to assess participant's overall impression of disease severity during the past 7 days with a 5-level scale of no symptoms, mild, moderate, severe or very severe. Data are reported for the percentage of participants with a PGID response of "No symptoms" at the specified timepoints.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 104
percentage of participants
  Week 2: number analyzed (Participants) | 101
  Week 2 | 4.0
  Week 4: number analyzed (Participants) | 100
  Week 4 | 4.0
  Week 8: number analyzed (Participants) | 96
  Week 8 | 14.6
  Week 12: number analyzed (Participants) | 90
  Week 12 | 10.0
  Week 16: number analyzed (Participants) | 92
  Week 16 | 12.0
  Week 20: number analyzed (Participants) | 84
  Week 20 | 14.3
  Week 24: number analyzed (Participants) | 80
  Week 24 | 23.8

21. Secondary Outcome: Percentage of Participants With PGID Response as No Symptoms or Mild Symptoms
Description: PGID is a single 1-item questionnaire designed to assess participant's overall impression of disease severity during the past 7 days with a 5-level scale of no symptoms, mild, moderate, severe or very severe. Data are reported for the percentage of participants with a PGID response of "No symptoms" or "Mild symptoms" at the specified timepoints.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 104
percentage of participants
  Week 2: number analyzed (Participants) | 101
  Week 2 | 26.7
  Week 4: number analyzed (Participants) | 100
  Week 4 | 46.0
  Week 8: number analyzed (Participants) | 96
  Week 8 | 59.4
  Week 12: number analyzed (Participants) | 90
  Week 12 | 65.6
  Week 16: number analyzed (Participants) | 92
  Week 16 | 68.5
  Week 20: number analyzed (Participants) | 84
  Week 20 | 64.3
  Week 24: number analyzed (Participants) | 80
  Week 24 | 67.5

22. Secondary Outcome: Percentage of Participants Who Rated Their Eczema Symptoms in the Patient Global Impression of Change (PGIC) as "Much Better"
Description: The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change in eczema symptoms since starting treatment as rated on a 7-point Likert scale anchored by (1) "much better" to (7) "much worse", with (4) = "no change". Data are reported for the percentage of participants who rated their eczema symptoms as "Much better" at the specified timepoints.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 114
percentage of participants
  Week 2 | 15.8
  Week 4 | 23.7
  Week 8: number analyzed (Participants) | 111
  Week 8 | 44.1
  Week 12: number analyzed (Participants) | 103
  Week 12 | 45.6
  Week 16: number analyzed (Participants) | 105
  Week 16 | 50.5
  Week 20: number analyzed (Participants) | 96
  Week 20 | 55.2
  Week 24: number analyzed (Participants) | 91
  Week 24 | 53.8

23. Secondary Outcome: Percentage of Participants Who Rated Their Eczema Symptoms in the PGIC as "Moderately Better"
Description: The PGIC is a single-item questionnaire designed to assess the participant's overall sense of whether there has been a change in eczema symptoms since starting treatment as rated on a 7-point Likert scale anchored by (1) "much better" to (7) "much worse", with (4) = "no change". Data are reported for the percentage of participants who rated their eczema symptoms as "Moderately better" at the specified timepoints.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 114
percentage of participants
  Week 2 | 14.0
  Week 4 | 27.2
  Week 8: number analyzed (Participants) | 111
  Week 8 | 23.4
  Week 12: number analyzed (Participants) | 103
  Week 12 | 28.2
  Week 16: number analyzed (Participants) | 105
  Week 16 | 27.6
  Week 20: number analyzed (Participants) | 96
  Week 20 | 25.0
  Week 24: number analyzed (Participants) | 91
  Week 24 | 23.1

24. Secondary Outcome: Number of Participants With Non-herpetic Skin Infection Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any untoward medical occurrence in a participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Data are reported for the number of participants with non-herpetic skin infection TEAEs. A summary of all serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 through Week 24
Population: Safety Set: All participants who were enrolled in the study and received at least 1 dose of dupilumab during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 124
Participants | 1

25. Secondary Outcome: Change From Baseline in Total Immunoglobulin (E) IgE
Description: Serum samples were collected to measure concentrations of IgE.
Time Frame: Weeks 4, 12 and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: kU/L
Arm/Group | Dupilumab
Number analyzed (Participants) | 107
kU/L
  Week 4 | -493.277 (1964.991)
  Week 12: number analyzed (Participants) | 105
  Week 12 | -2284.021 (5579.402)
  Week 24: number analyzed (Participants) | 87
  Week 24 | -3177.471 (6959.014)

26. Secondary Outcome: Percent Change From Baseline in Total IgE
Description: Serum samples were collected to measure concentrations of IgE.
Time Frame: Weeks 4, 12 and 24
Population: Here 'n' = Number of evaluable participants at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Dupilumab
Number analyzed (Participants) | 115
percent change
  Week 4: number analyzed (Participants) | 107
  Week 4 | -6.277 (62.301)
  Week 12: number analyzed (Participants) | 105
  Week 12 | -39.703 (25.145)
  Week 24: number analyzed (Participants) | 87
  Week 24 | -50.375 (69.291)

27. Secondary Outcome: Trough Concentration of Functional Dupilumab in Serum
Description: Adolescents and adults received 1 of 2 dose regimens based on age and body weight. The trough concentration of functional dupilumab in serum for the 2 dose regimens at the specified time points are presented. Participants treated and had at least one evaluable post-first-dose concentration measurement.
Time Frame: Week 12 and Week 24
Population: Pharmacokinetic (PK) Analysis Set: All participants who received any study drug and who had at least 1 non-missing PK result following the first dose of any study drug. Analysis was based on the treatment received. Overall number of participants analyzed = participants evaluable for the outcome measure. Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Dupilumab
Number analyzed (Participants) | 114
mg/L
  Dose Regimen 1: Week 12: number analyzed (Participants) | 5
  Dose Regimen 1: Week 12 | 40.8 (28.7)
  Dose Regimen 2: Week 12: number analyzed (Participants) | 104
  Dose Regimen 2: Week 12 | 43.9 (28.4)
  Dose Regimen 1: Week 24: number analyzed (Participants) | 6
  Dose Regimen 1: Week 24 | 43.9 (28.0)
  Dose Regimen 2: Week 24: number analyzed (Participants) | 84
  Dose Regimen 2: Week 24 | 49.6 (33.4)

28. Primary Outcome: Percentage of Participants With ≥75% Reduction From Baseline in Eczema Area and Severity Index (EASI) Score (EASI-75)
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 24.
Time Frame: Week 24
Population: Here 'n' = number of evaluable participants at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dupilumab
Number analyzed (Participants) | 100
percentage of participants | 76.0 [66.43 to 83.98]

ADVERSE EVENTS:
Time Frame: Day 1 through Week 24
Description: Safety Set: all participants who were enrolled in the study and received at least 1 dose of dupilumab during the study.
Arm/Group | Dupilumab
All-Cause Mortality (participants affected / at risk) | 1/124
Serious Adverse Events (participants affected / at risk) | 7/124
Other Adverse Events (participants affected / at risk) | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dupilumab (N=124)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Intussusception (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05590585/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT05590585/SAP_001.pdf